CLINICAL TRIAL: NCT06215183
Title: The Effect of Music on Pain, Anxiety and Satisfaction During Intrauterine Device Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sümeyye Köse (Other)
Responsible Party: Sponsor-Investigator, Sümeyye Köse, Phd Student, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SKOSE
Record Dates: First submitted 2024-01-07; First posted 2024-01-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Reproductive Health; Pain; Women Health
Keywords: Intrauterine device; Pain; Anxiety; Satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial.
Who Masked: Participant
Masking Description: The evaluation was made by the participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Women in the intervention group applying for IUD application will listen to music for 5 minutes before, during and after the procedure.
  Interventions: Other: Music therapy
- Control Group (No Intervention): Women in the control group applying for IUD application will not be subjected to any intervention other than routine IUD insertion procedures.

INTERVENTIONS:
Other: Music therapy — Women applying for IUD application will receive music therapy for 5 minutes before the procedure, during the IUD application, and for 5 minutes after the procedure.
  Arms: Intervention Group

SUMMARY:
This study was planned to determine the effect of music listened to during intrauterine device application on pain,anxiety and satisfaction.

DETAILED DESCRIPTION:
The randomized controlled and experimental study will be conducted with 70 women who apply to a Maternal and Child Health and Family Planning Center to have an Intrauterine Device (IUD). Women in the experimental group (n=35) will listen to music before, during and after the IUD application process, and the control group (n=35) will undergo routine IUD application. Information Form containing sociodemographic information, Situational Anxiety

ELIGIBILITY:
Inclusion Criteria:

* Knowing how to read and write,
* Not having had an IUD inserted before,
* Being between the ages of 18-49,
* No hearing-related problems,
* Not having used analgesic or anesthetic medication within 24 hours before or during the procedure,
* Voluntarily participating in the study,

Exclusion Criteria:

* The woman has a cognitive and auditory problem
* Having a history of cervical surgery

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 30 minütes
  Data will be collected using the State Anxiety Inventory. The answer options collected in four classes on the State Anxiety Inventory scale are: (1) Not at all, (2) A little, (3) A lot and (4) Completely; The options on the trait anxiety scale are (1) Rarel, (2) Sometimes, (3) A lot of the time, and (4) Almost always. The higher the score obtained from the scales, the higher the person's anxiety is. The total score obtained from the scale varies between 20-80, and 20-39 indicates a mild anxiety level, 40-59 indicates a medium anxiety level, 60-79 indicates a high anxiety level, and 80 points indicates a panic anxiety level.
Pain Level | 30 minütes
  Data will be collected using the Visual Analogue Scale. Pain can be given a score between 0 and 10 on the scale.The higher the scale score, the greater the pain.

SECONDARY OUTCOMES:
Satisfaction Level | 30 minütes
  Data will be collected using the Visual Analog Scale. Satisfaction can be given a score between 0 and 10 on the scale. The higher the scale score, the higher the satisfaction level.

CONTACTS AND LOCATIONS:
Locations (1):
- Pendik District Health Directorate Maternal Child Health and Family Planning Center, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No